CLINICAL TRIAL: NCT06123546
Title: Effectiveness of a Patient-oriented Discharge Summary for Older Inpatients Discharged Home.
Brief Title: Effectiveness of a Patient-oriented Discharge Summary
Acronym: PODS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Dr. Sc. Cedric Mabire, RN PhD, Associate Professor, University of Lausanne
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PODS_2024
Record Dates: First submitted 2023-07-05; First posted 2023-11-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Multimorbidity

STUDY DESIGN:
Intervention Model Description: Months 1-4: recruitment/data collection of the control group Month 5: implementation of the intervention Month 5-8: recruitment/data collection of the intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual discharge preparation (No Intervention): Discharge teaching according to the usual discharge preparation process in participating units
- Teaching with a patient-oriented discharge summary (Experimental): Discharge teaching with a patient-oriented discharge summary, using the teach-back technique and inclusion of caregivers
  Interventions: Other: Patient oriented discharge summary

INTERVENTIONS:
Other: Patient oriented discharge summary — The intervention consists of three components: the patient-oriented discharge summary (PODS), the teach-back technique and the involvement of caregivers.
  The PODS will be completed with participants over the course of the hospitalisation as teaching content related to the six sections of information is delivered. Participants will take the PODS home at discharge to use it as a reference for relevant and individualized discharge information in the post-discharge period.
  Healthcare providers will receive a training refresher on the teach-back technique and will be reminded to use it when they deliver discharge teaching during participants' hospital stay.
  Involvement of caregivers will include early identification by the healthcare provider responsible for patient admission of a caregiver who will provide care at home, at least one teaching session during hospitalization and the review of the PODS the day of discharge.
  Other Names: PODS
  Arms: Teaching with a patient-oriented discharge summary

SUMMARY:
The discharge preparation is a difficult time to provide teaching, as older patients and their caregivers are often overwhelmed by a substantial amount of information and stressed about leaving hospital. As a result, 40-80% of patients forget or remember incorrectly the information discussed during hospitalisation, resulting in unmet needs, poor adherence to postdischarge care and increased use of health care services in the postdischarge period. The Patient-Oriented Discharge Summary (PODS) is a simple, one-page tool to be completed with key information, such as the reason for hospitalisation, warning signs to look out for, contact information, treatment plan and upcoming medical appointments. The PODS study will assess the effectiveness of the PODS on the quality of the transition between hospital and patients' home and problems and unmet needs after discharge.

DETAILED DESCRIPTION:
Full Title: The effectiveness of a patient-oriented discharge summary for older inpatients discharged home Primary objective: To evaluate the effectiveness of a patient-oriented discharge summary on the quality of care transition for older patients discharged home Secondary objective: To evaluate the effectiveness of a patient-oriented discharge summary on caregivers' perceived self-efficacy in the transition and older patients' problems and unmet needs after hospitalization.

Hypothesis are that:

H1. Patients exposed to the PODS, compared with patients receiving usual discharge preparation, would have improved quality of care transition H2. Patients exposed to the PODS, compared with patients receiving usual discharge preparation, would have less problems and unmet needs during the postdischarge period, including 7-days readmission and unplanned use of healthcare services H3. Caregivers of patients exposed to the PODS would have improved perceived self-efficacy in the transition compared to patients receiving usual discharge preparation

Study design: This monocentric study has a quasi-experimental design, using a non-randomised 2 group pre/post-intervention comparative design. This design was chosen to provide preliminary evidence on the effectiveness of the proposed intervention. As the implementation of evidence-based interventions is a major objective of health care services, this pilot study is prerequisite for judging the relevance and evaluate if the patient-oriented discharge summary is likely to be effective for a future randomized clinical study. The recruitment period is planned for 8 months. Project duration for each patient will correspond to the duration between recruitment day and 5-7 days post-discharge.

Study intervention:

The intervention consists of three components: the patient-oriented discharge summary, the teach-back technique and the involvement of caregivers. The healthcare team of participating units will be trained in the intervention components.

The patient-oriented discharge summary is individualized discharge tool, containing meaningful information for patients presented in an easy-to-understand format. This one-page document contains six sections of information to be completed by the healthcare team: 1.) reason for hospitalization, 2.) medications, 3.) warning signs and symptoms to watch out, 4.) changes to daily activities and health behaviors, 5.) upcoming follow-up appointments and 6.) contact information. The nurse responsible for hospital admission will print and give a PODS to the participant and explain the purpose of the document. The PODS will be kept in the participants' room during the hospital stay. In each study unit, a "PODS champion" encourage the healthcare team to help and encourage patients to fill out the PODS over the course of the hospitalisation as teaching content related to the six sections of information occurs. The day of discharge, the physician responsible for participants' hospital discharge will review and verify that the information written in the PODS correspond to the teaching content that was discussed. Participants will take the PODS home at discharge to use it as a reference for relevant and individualized discharge information in the post-discharge period.

The second component of the intervention is the use of the teach-back technique, as an evidence-based approach to confirm the full comprehension of teaching content. The teach-back consist in asking patients to repeat what they have understood in their own words. Healthcare providers will receive a training refresher on the teach-back technique and will be reminded to use it when they deliver discharge teaching during participants' hospital stay.

The third component is the involvement of caregivers in the discharge teaching. This will include early identification by the healthcare provider responsible for patient admission of a caregiver who will provide care at home, at least one teaching session during hospitalization and the review of the PODS the day of discharge. The importance of caregiver involvement will be emphasized to healthcare providers in the training session.

Intervention procedure:

To reduce potential performance bias, the healthcare teams of the units will attend a one-hour training session in the intervention. The training will include and adapt the training resources made available by the PODS developers (https://pods-toolkit.uhnopenlab.ca/resources/#resources-train). Content of the training session will include an introduction about the PODS, and guidance on how to fill in the tool and use the teach-back technique. A short video clip will also be available to summarize key information regarding the PODS. Training sessions will be conducted at the end of the control phase to prevent contamination. A training refresher will be provided to the healthcare team twice a month during the intervention phase. Weekly meetings will be conducted by the investigator with the healthcare teams in the units to ensure that procedures have been carried out correctly. If the healthcare teams have any questions during the intervention phase, they can contact the research team at anytime.

After giving informed consent, the intervention begins by the identification by the healthcare provider responsible for patient admission of a caregiver who will provide care at home. Participants will receive the PODS with explanations about how it will be used during the hospital stay. The PODS will remain in the patient's room as it will be used as a support for the discharge teaching. The healthcare teams will provide the discharge teaching according to the description of the intervention (see 2.4) during the hospital stay. The day of discharge, the content of the PODS will be verified by the physician and the healthcare provider responsible for discharge or the liaison nurse (to be defined by the units) will inform the home care services that the participant is discharged with this summary.

Recruitment, screening and informed consent procedure:

A convenience sample of patient participants will be recruited in two participating units of a regional Swiss hospital. Recruitment will occur upon patient admission. In each unit, 21 control patients will be recruited during the pre-implementation phase of the intervention. This recruitment will last approximately four months. After this control period, 21 other patients will be recruited to receive the intervention.

For the control and the intervention groups, newly admitted inpatients will be routinely screened for eligibility in the two units by project coordinators. Project coordinators will be healthcare professionals of the study units, responsible for the study coordination at the hospital. They will be trained on participants inclusion criteria and inform the research collaborator of eligible patients and caregivers. The research collaborator will be trained by the investigator on informed consent and providing information to ensure patients' understanding, and ethical and responsible conduct of research. The research collaborator will approach the patient to discuss the study at the most appropriate time as deemed by them (outside of the time for care or treatment). The research collaborator will explain to each participant the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits and any discomfort it may entail. Participants will be informed that the participation in the study is voluntary and that they may withdraw from the study at any time and that withdrawal of consent will not affect their subsequent medical assistance and treatment. Patient participants will be informed that their medical records may be examined by authorised individuals other than their treating physician. Eligible patients will also be invited to participate to postdischarge interviews, additionally to the data collection with questionnaires (CTM-15). They will be informed that interviews will be audiotaped.

All participants for the study will be provided a participant information sheet and a consent form describing the study and providing sufficient information for participant to make an informed decision about their participation in the study. Participants will have a 24-hour reflection period and the investigator will remain available, including by telephone, for any questions. The formal consent of a participant, using the approved consent form, will be obtained before the participant is submitted to any study procedure. The consent form will be signed and dated by the investigator or his designee at the same time as the participant sign. A copy of the signed informed consent will be given to the study participant. The consent form will be retained as part of the study records.

When there is an identified caregiver for the participant, the caregiver will be approached at the most opportune time, preferably in the presence of the concerned patient. The research collaborator will inform the caregiver of the study and its implication for the patient participant. Caregivers who consent to participate will sign a consent form. Their participation will consist of completing the FACT questionnaire and, as an option, taking part in the interview 5-7 days after patients' discharge.

Data collection procedure:

A research collaborator will be responsible for collecting the data and administering the questionnaires. The investigator will train the research collaborator on the protocol (in particular eligibility criteria, ethical consideration related to participant information and consent, conducting interviews, questionnaire administration, scoring and data recording to limit the risk of measure bias. Weekly meetings will be conducted by the investigator with the research collaborator to ensure that procedures have been carried out correctly.

After giving informed consent, the research collaborator will ask participants to complete the baseline data form and will collect data from Electronic Health Record. During the hospital stay, the project coordinators on sites will inform the research collaborator of participants' planned discharge day. The day of discharge or the day before, the research collaborator will visit the participant to plan the phone call or the home visit (according to their preferences) 5-7 days later to collect patients and caregivers' outcomes. Interviews with participating dyads or patients only will also be scheduled. Five to seven days after discharge, the investigator will support participants in completing the CTM-15 and the FACT tool. Interviews will be conducted following the interview guide and recorded. If participants raise a major problem at home during interviews that would be necessary to be solved for the participants' safety, the investigator will ask the agreement of participants to notify their physician in the community.

ELIGIBILITY:
Inclusion criteria:

* Being discharged home
* Able to speak, read and write in French
* Being hospitalized for more than 48H in participating medical units
* Being able to give informed consent as documented by signature

Exclusion criteria:

• Inability to follow the procedures of the study according to the health care team, due to language problems or cognitive impairment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Quality of care transition measured with the Care Transition Measure Tool (CTM-15) | 5-7 days after discharge
  Quality of care transition will be measured by the Care Transition Measure Tool (CTM-15) at 5-7 days post-discharge. The CTM is a 15-item self-report questionnaire to evaluate the quality of the posthospital care transition experience from patient's perspective, in four factors: critical understanding, preferences important, management preparation, care plan. Responses for each item range from 1 = ''strongly disagree,'' to 4 = "strongly agree". A mean score is calculated by adding the value of each responded item ad divide this score by the number of answered items. The score is converted on a 0-100 scale using the formula: ((mean score - 1)/3)*100. Cronbach's alpha for the CTM-15 is 0.93. Construct validity showed that CTM scores had a small negative correlation with age (r = -0.16, p = 0.03 and length of stay (r = 0.14, p = 0.05).

SECONDARY OUTCOMES:
Family Caregiver Activation in Transitions (FCAT) | 5-7 days after discharge
  Perceived caregivers self-efficacy with respect to transition-specific tasks will be measured with the Family Caregiver Activation in Transitions (FCAT) Tool at 5-7 days post-discharge. The FCAT is a 10-item self-report questionnaire, exploring with responses ranging from 1 = "Disagree strongly" to 6 = "Agree strongly". Psychometric testing showed that the items function as a unidimensional construct, with an estimated person-separation reliability of 0.84 .
Problems and unmet needs experienced during the week after discharge | 5-7 days after discharge
  Problems and unmet needs will be collected during interviews with 15-18 patient participants and 5-8 caregivers 5 to 7 days after discharge. The participants will be asked open-ended questions on post-discharge problems and unmet needs, using the photolanguage technique. Participants will be given a selection of pictures representing common difficulties experiences by older patients. They will be encouraged to choose images that resonate with their experiences, thoughts, and emotions following discharge. Through this visual dialogue, the research collaborator will support participants to express their concerns, and challenges in transitioning back to independent living or adjusting to new caregiving arrangements. By using photographs as a medium, photolanguage

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de Morges, Morges, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Pellet J, Solano Araujo R, Kathirkamu S, Hilfiker R, Bartholdi N, Mabire C. Implementing a patient-oriented discharge summary to improve hospital-to-home transitions in older adults: lessons from a hybrid study. Front Health Serv. 2026 Jan 16;5:1730127. doi: 10.3389/frhs.2025.1730127. eCollection 2025. PMID 41623518